CLINICAL TRIAL: NCT03339232
Title: BCAA Supplemental Study: Branched Chain Amino Acid and Physical Activity to Improve Muscle Mass in Patients With Cirrhosis
Brief Title: BCAA Supplemental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Eric Kallwitz, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 210050
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of three arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Participants will receive standardized information about a healthy diet, including the potential benefit of small, frequent meals and nighttime snacking . In addition, the treating hepatologist will counsel participants on the benefits of increased physical activity. These recommendations will be provided at the beginning of the study. The usual care arm reflects current clinical practice. Participants will be asked to keep an exercise log detailing type and duration of at home physical activity.
- BCAA Supplement (Other): BCAA powder (Bulk Supplements®) will be provided as the powder was found to be easier to swallow. Each teaspoon contains 1788 mg of BCAA and participants will take 7 teaspoons (12.5 grams of BCAA) per day divided into three separate servings. Each teaspoon contains L-leucine, isoleucine and valine in a 2:1:1 ratio. BCAA will be provided by the study investigators and half will be provided at baseline study visit and the second half at the week 6 visit. In addition, the treating hepatologist will provide standardized information about the potential benefits of small, frequent meals, nighttime snacking and increased physical activity at the beginning of the study. Participants will be asked to keep an exercise log detailing type and duration of at home physical activity.
  Interventions: Dietary Supplement: BCAA Supplement
- BCAA supplement plus supervised physical activity (Other): BCAA supplement will be as described for group 2, above. Study coordinators will supervise the physical activity program for study participants at the Loyola Fitness Center. Participants will attend the fitness center one hour each week; the fitness session will consist of low-impact aerobic physical activity, beginning with walking on the indoor track and possibly building to a recumbent exercise bicycle and light resistance training. Participants will be given a list of exercises to perform at home at least two times during the week with a goal of >90 minutes of physical activity per week. Participants will be asked to keep an exercise log detailing type and duration of at home physical activity which they will return during the weekly fitness center sessions. In addition, the treating hepatologist will provide standardized information about the potential benefits of small, frequent meals, nighttime snacking and increased physical activity at the beginning of the study.
  Interventions: Dietary Supplement: BCAA Supplement; Other: Physical Activity

INTERVENTIONS:
Dietary Supplement: BCAA Supplement — Each teaspoon contains 1788 mg of BCAA and participants will take 7 teaspoons (12.5 grams of BCAA) per day divided into three separate servings. Each teaspoon contains L-leucine, isoleucine and valine in a 2:1:1 ratio.
  Arms: BCAA Supplement; BCAA supplement plus supervised physical activity
Other: Physical Activity — Supervised low impact aerobic physical activity for one hour each week.
  Arms: BCAA supplement plus supervised physical activity

SUMMARY:
The central hypothesis of this study is that BCAA supplementation and BCAA supplementation plus low-intensity activity will improve muscle mass and HRQOL in cirrhotic patients compared to usual care

DETAILED DESCRIPTION:
The purpose of this study is to look at the impact of including a physical activity program and/or a nutritional supplement along with your regular care. The nutritional supplement used in this study consists of branched-chain amino acids (BCAAs). BCAAs are found in certain foods and are readily available as dietary supplements.

The investigators in this study will look at how the physical activity and nutritional supplement program might affect patients' health outcomes, and if this program can maintain or even increase muscle mass in patients with cirrhosis.

Participants will be randomized in three groups:

1. Standard Care: If the participant is randomized to this group, they will receive the same medical care for their cirrhosis as they would if they were not participating in the study. The doctor will provide them with some general information about healthy diet and exercise. They will also be asked to keep an exercise log of the type of physical activity they do on your own.
2. Nutritional Supplement: BCAAs: If the participant is randomized to this group, they will be provided with BCAA powder to take during the 12 weeks of the study. They will be asked to take 7 teaspoons per day. They will take 2-3 teaspoons after each meal. The doctor will also provide them with some general information about healthy diet and exercise, and they will also be asked to keep an exercise log of any physical activity they do on your own.
3. Nutritional Supplement and Supervised Physical Activity: If the participant is randomized to this group, they will be provided with BCAA powder and be asked to participate in one hour per week of supervised fitness instruction at the Loyola Center for Fitness. The fitness instruction will consist of low-impact aerobic exercise such as walking or riding an exercise bicycle. They will also be given a list of exercises to perform at home at least two times during the week and be asked to keep an exercise log of their physical activity. The doctor will provide them with some general information about healthy diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis with ascites
2. MELD-Na score<25

Exclusion Criteria:

1. Pregnancy
2. Inability to engage in low-intensity physical activity due to any condition
3. Active acknowledged alcohol or substance abuse
4. Inability to complete protocol assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Muscle Mass | 12 weeks
  Appendicular lean muscle mass will be measured by whole body DXA using a standard protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scaglione S, Kliethermes S, Cao G, Shoham D, Durazo R, Luke A, Volk ML. The Epidemiology of Cirrhosis in the United States: A Population-based Study. J Clin Gastroenterol. 2015 Sep;49(8):690-6. doi: 10.1097/MCG.0000000000000208. PMID 25291348
- [Background] Alter MJ, Kruszon-Moran D, Nainan OV, McQuillan GM, Gao F, Moyer LA, Kaslow RA, Margolis HS. The prevalence of hepatitis C virus infection in the United States, 1988 through 1994. N Engl J Med. 1999 Aug 19;341(8):556-62. doi: 10.1056/NEJM199908193410802. PMID 10451460
- [Background] Browning JD, Szczepaniak LS, Dobbins R, Nuremberg P, Horton JD, Cohen JC, Grundy SM, Hobbs HH. Prevalence of hepatic steatosis in an urban population in the United States: impact of ethnicity. Hepatology. 2004 Dec;40(6):1387-95. doi: 10.1002/hep.20466. PMID 15565570
- [Background] Kallwitz ER, Guzman G, TenCate V, Vitello J, Layden-Almer J, Berkes J, Patel R, Layden TJ, Cotler SJ. The histologic spectrum of liver disease in African-American, non-Hispanic white, and Hispanic obesity surgery patients. Am J Gastroenterol. 2009 Jan;104(1):64-9. doi: 10.1038/ajg.2008.12. PMID 19098851
- [Background] Darmon N, Drewnowski A. Does social class predict diet quality? Am J Clin Nutr. 2008 May;87(5):1107-17. doi: 10.1093/ajcn/87.5.1107. PMID 18469226
- [Background] Gordon-Larsen P, Nelson MC, Page P, Popkin BM. Inequality in the built environment underlies key health disparities in physical activity and obesity. Pediatrics. 2006 Feb;117(2):417-24. doi: 10.1542/peds.2005-0058. PMID 16452361
- [Background] Merli M, Giusto M, Gentili F, Novelli G, Ferretti G, Riggio O, Corradini SG, Siciliano M, Farcomeni A, Attili AF, Berloco P, Rossi M. Nutritional status: its influence on the outcome of patients undergoing liver transplantation. Liver Int. 2010 Feb;30(2):208-14. doi: 10.1111/j.1478-3231.2009.02135.x. Epub 2009 Oct 14. PMID 19840246
- [Background] Hong HC, Hwang SY, Choi HY, Yoo HJ, Seo JA, Kim SG, Kim NH, Baik SH, Choi DS, Choi KM. Relationship between sarcopenia and nonalcoholic fatty liver disease: the Korean Sarcopenic Obesity Study. Hepatology. 2014 May;59(5):1772-8. doi: 10.1002/hep.26716. Epub 2014 Mar 24. PMID 23996808
- [Background] Issa D, Alkhouri N, Tsien C, Shah S, Lopez R, McCullough A, Dasarathy S. Presence of sarcopenia (muscle wasting) in patients with nonalcoholic steatohepatitis. Hepatology. 2014 Jul;60(1):428-9. doi: 10.1002/hep.26908. Epub 2014 May 27. No abstract available. PMID 24990106
- [Background] Hayashi F, Matsumoto Y, Momoki C, Yuikawa M, Okada G, Hamakawa E, Kawamura E, Hagihara A, Toyama M, Fujii H, Kobayashi S, Iwai S, Morikawa H, Enomoto M, Tamori A, Kawada N, Habu D. Physical inactivity and insufficient dietary intake are associated with the frequency of sarcopenia in patients with compensated viral liver cirrhosis. Hepatol Res. 2013 Dec;43(12):1264-75. doi: 10.1111/hepr.12085. Epub 2013 Mar 12. PMID 23489325